CLINICAL TRIAL: NCT01415557
Title: The Effects of Regular Consumption of a Multiple Micronutrient Fortified Beverage on the Micronutrient Status of Indian Schoolchildren and on Their Mental and Physical Performance
Brief Title: Effect of Regular Consumption of Micronutrient Fortified Beverage on the Micronutrient Status of Indian Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KFTSJRI2011
Record Dates: First submitted 2011-07-22; First posted 2011-08-12 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: micronutrient; healthy children; vitamins; minerals; cognition; physical performance; iron; Micronutrient status; Cognitive Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Fortified Control Product (Placebo Comparator): Non-fortified control beverage
  Interventions: Other: Non-Fortified Control Product
- Micronutrient Fortified Test Product (Active Comparator): Micronutrient fortified test beverage
  Interventions: Other: Micronutrient Fortified Test Product

INTERVENTIONS:
Other: Non-Fortified Control Product — Non-Fortified Control Beverage
  Arms: Non-Fortified Control Product
Other: Micronutrient Fortified Test Product — Micronutrient Fortified Test Beverage
  Arms: Micronutrient Fortified Test Product

SUMMARY:
The purpose of this study is to assess the impact of regular consumption of micronutrient fortified drink in improving nutritional and micronutrient status in Indian school children. The test beverage will be fortified with both, vitamins and minerals.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy school going children
* not severely malnourished weight-for-height z-score ≥-2 not severely anemic (Hb<8g/dl)
* Age: 7-10 years
* Not taking any food supplements/fortified drinks
* Not planning to move out during the study duration

Exclusion Criteria:

* Age: <7 and >10 years
* Severe anemia (Hb < 8 g/dl)
* Severely malnourished children with weight-for-height z-score <-3 will be excluded.
* Cardiovascular disease on clinical examination or history
* Underlying respiratory disease with impairment of lung function
* Physical disability which can interfere or limit performance of tests
* Recent history (3 months prior) of serious infections, injuries and/ or surgeries
* Any food allergy or food intolerance
* Participation in any nutritional study in the last 1year
* Children consuming nutritional supplements and/ or health food drinks

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 227 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the micronutrient status in the study subjects at 6 months | 6 months
  The primary outcome measures will be change from baseline in the micronutrient status in the study subjects at end of intervention.

SECONDARY OUTCOMES:
Change from baseline in cognitive performance at 6 months | 6 months
  Change from baseline in cognitive test scores at the end of the intervention for all subjects.
Change from baseline in the physical performance at 6 months | 6 months
  Change from baseline in the physical test scores at end of intervention for all subjects
Change from baseline in the fatigue score at 6 months | Baseline and Endline (six months)
  Change from baseline in the fatigue score at end of intervention for all subjects
Morbidity Assessment | 6 months
  Morbidity will be recorded on a weekly basis from the start until the end of the intervention
Prevalence of Micronutrient Deficiency | 6 months
  Prevalence of micronutrient deficiency in each study arm at the end the intervention
Change from baseline in anthropometric scores at 6 months | 6 months
  Change from baseline in anthropometric measures (Standardized (WHO, 2007) weight for age, height for age and BMI for age of the study subjects) at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Prashanth Thankachan, PhD, Principal Investigator — St. John's Research Institute
Locations (1):
- St. Johns Research Institute, Bangalore, Karnataka, India

REFERENCES:
- [Derived] Kuriyan R, Thankachan P, Selvam S, Pauline M, Srinivasan K, Kamath-Jha S, Vinoy S, Misra S, Finnegan Y, Kurpad AV. The effects of regular consumption of a multiple micronutrient fortified milk beverage on the micronutrient status of school children and on their mental and physical performance. Clin Nutr. 2016 Feb;35(1):190-198. doi: 10.1016/j.clnu.2015.02.001. Epub 2015 Feb 21. PMID 25746819